CLINICAL TRIAL: NCT02943928
Title: Placement of the Double-Lumen Tube Without Fiberoptic Bronchoscope Assistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2016A123
Record Dates: First submitted 2016-10-23; First posted 2016-10-25 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Therapeutic Procedural Complication
MeSH Terms: interventions — Laryngoscopes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laryngoscope and chest CT image (Experimental): First,the operator calculate the distance between the carina and the glottis by CT image and make s marker on the double lumen endotracheal tube. Then the operator when inserted into the double lumen tube under the visualof laryngoscope until see marker just at the glottis.
  Interventions: Device: laryngoscope and chest CT image
- Traditional method by experience (Experimental): Operator inserted the double lumen tube by experience
  Interventions: Device: traditional method by experience

INTERVENTIONS:
Device: laryngoscope and chest CT image — First,the operator calculate the distance between the carina and the glottis by CT image and make s marker on the double lumen endotracheal tube. Then the operator when inserted into the double lumen tube under the visualof laryngoscope until see marker just at the glottis
  Arms: laryngoscope and chest CT image
Device: traditional method by experience — Operator inserted the double lumen tube by experience
  Arms: Traditional method by experience

SUMMARY:
laryngoscope combined with chest CT in double lumen endotracheal tube accurate positioning

DETAILED DESCRIPTION:
Comparing the traditional method of double lumen endotracheal tube intubation and laryngoscope combined with chest CT guide the precise localization of double lumen endotracheal tube

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 35 kg/m2
* ASA classifications of I-III, modified Mallampati classification 1 or 2 general anesthesia were included-

Exclusion Criteria:

* Exclusion criteria included age younger than 18 yr
* ASA class IV or V
* Abnormalities of the heart, brain, liver, lung, kidney and coagulation functions-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Intubation Time | Ten minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ximing Qi, Study Director — The First Hospital of Qinhuangdao
Locations (1):
- 中国, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes